CLINICAL TRIAL: NCT03203187
Title: The Effect of Daily Mango Intake (Mangifera Indica L.) on Cardiovascular Health
Brief Title: The Effect of Daily Mango Intake on Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 894860
Record Dates: First submitted 2017-02-27; First posted 2017-06-29 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No mango intake (Placebo Comparator): No mango intake for two weeks
  Interventions: Other: No intervention
- 330 grams of daily mango intake (Experimental): 330 grams (2 cups) of daily mango intake for two weeks
  Interventions: Other: Mango

INTERVENTIONS:
Other: Mango — 330 grams (2 cups) of daily mango intake for two weeks, one cup in the morning, the other in the evening
  Arms: 330 grams of daily mango intake
Other: No intervention — No mango intake for two weeks.
  Arms: No mango intake

SUMMARY:
In the current proposal the investigators seek to evaluate the acute and short-term effects of mango intake on vascular and platelet function in postmenopausal women between 50 and 70 years old.

Our aims are 1) to determine if two weeks of daily mango intake will result in favorable changes in measures of vascular function, as measured using peripheral arterial tonometry (PAT) and platelet reactivity, in overweight and obese postmenopausal women. 2) to determine if two weeks of daily mango intake will change the fermentation capacity of gut microbiota.

Investigators hypothesize that the daily intake of 330 grams of mango (2 cups) will significantly increase PAT while reducing platelet aggregation after 2 hours and two weeks of daily intake.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female: 50-70 years
* Women: lack of menses for at least one year and FSH 23-116.3 mlU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing participate in all study procedures
* BMI 25.0 - 40 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* BMI ≥ 40 kg/m2
* Dislike or allergy for mango
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Alcohol consumption > 3 drinks/week (i.e. 1 bottle of beer, ½ glass of wine, and 1 shot of hard liquor)
* Fruit consumption ≥ 2 cups/day
* Vegetable consumption ≥ 3 cups/day for females
* Fatty Fish ≥ 3 times/week
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and Stroke
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Liver, CBC or Chemistry panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Currently taking prescription drugs or supplements, other than thyroid medication.
* Use of multi-vitamin and mineral other than a general formula of vitamins and minerals that meet the RDA
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Screening LDL ≥ 190 mg/dl for those who have 0-1 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].

(using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp);

* Screening LDL ≥ 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL], and a Framingham 10-year Risk Score 10-20% (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp).
* Current enrollee in a clinical research study.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-02 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Acute vascular function | change from baseline to 2 hours compared on days 0 14 and 28
  Comparison of the effect of mango on acute vascular function between baseline and 2-hour postprandial response using PAT.
Long-term vascular function | Comparison of day 0, 14, and 28
  The effect of mango on long-term vascular function between baseline, two week, and four week time points using PAT

SECONDARY OUTCOMES:
Acute platelet aggregation | change from baseline to 2 hours compared on days 0 14 and 28
  Comparison of the effect of mango on acute platelet aggregation between baseline and 2-hour postprandial time.
Long-term platelet aggregation | Comparison of day 0, 14, and 28
  Comparison of the effect of mango on long-term platelet aggregation baseline, two week, and four week time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Regal Human Nutrition Research Center, Davis, California, United States